CLINICAL TRIAL: NCT07195084
Title: A Phase I Clinical Study to Explore the Safety and Efficacy of Hypervision Proton Surgery (HyPROS) for Early-stage Non-small Cell Lung Cancer
Brief Title: To Explore the Safety and Efficacy of Hypervision Proton Surgery (HyPROS) for Early-stage Non-small Cell Lung Cancer
Acronym: HyPROS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Collaborators: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Shuanghu Yuan, Professor, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HyPROS
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; Hypervision proton surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton radiotherpy (Experimental): Proton radiotherapy 34GyE/f or 39GyE/f
  Interventions: Radiation: Hypervision proton surgery

INTERVENTIONS:
Radiation: Hypervision proton surgery — Proton radiaotherapy (34GyE or 39GyE)

SUMMARY:
This study was a single-center, single-arm clinical study to evaluate the safety and efficacy of hypervision proton surgery with single large fractionated doses (34GyE and 39GyE) in the treatment of early peripheral NSCLC.

DETAILED DESCRIPTION:
This study adopted a dose escalation protocol (an improved "two-stage two-dose group" design) to explore the safety and efficacy of visual proton surgery (single large fractionated doses of 34GyE and 39GyE) in the treatment of early peripheral NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years old
* Karnofsky Performance Status > 80
* NSCLC confirmed by cytology or histology
* Early-stage tumors are defined as T1 (≤3cm) N0M0 based on enhanced computed tomography (CT) and positron emission tomography (PET)
* The tumor must be more than 2 cm away from the proximal bronchial tree in all directions (the proximal bronchial tree is defined as 2 cm from the distal end of the trachea, the protrusion and the named lobar bronchus up to its first bifurcation)
* FEV1 ≥ 1 L, FEV1 ≥ 40% of the predicted value (either one is sufficient); DLCO ≥ 40% of the predicted value
* The patient can tolerate PET-CT examination
* For female study participants of childbearing age, the urine or serum pregnancy test was negative within 7 days prior to the first administration of the study drug. If the result of the urine pregnancy test is positive, a blood pregnancy test is required

Exclusion Criteria:

* Other malignant tumors occurred concurrently within 2 years before enrollment
* A history of chest radiotherapy in the past
* It is planned to use other anti-tumor treatments within the regimen treatment (within 4 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2027-09-19 (Estimated); Study Completion 2028-09-19 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade ≥ 3 psAEs at 1 month | 1 month after proton radiotherapy
  Radiation induced adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE)
The incidence of grade ≥ 3 psAEs at 1 year | 1 year after proton radiotherapy
  Radiation induced adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Primary tumor control at 1 year | 1 year after proton radiotherapy
  Primary tumor control at 1 year
Disease-free survival time | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Disease-free survival time
Overall survival time | From date of treatment until the date of death
  Overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Shuanghu Yuan, PhD, Principal Investigator — Anhui Provincial Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: A Randomized Phase 2 Study Comparing 2 Stereotactic Body Radiation Therapy Schedules for Medically Inoperable Patients With Stage I Peripheral Non-Small Cell Lung Cancer: NRG Oncology RTOG 0915 (NCCTG N0927) — https://pubmed.ncbi.nlm.nih.gov/26530743/
- See also: Long-term Follow-up on NRG Oncology RTOG 0915 (NCCTG N0927): A Randomized Phase 2 Study Comparing 2 Stereotactic Body Radiation Therapy Schedules for Medically Inoperable Patients With Stage I Peripheral Non-Small Cell Lung Cancer — https://pubmed.ncbi.nlm.nih.gov/30513377/